CLINICAL TRIAL: NCT00551369
Title: A Phase II Trial of Stereotactic Body Radiation Therapy (SBRT) in the Treatment of Patients With Operable Stage I/II Non-Small Cell Lung Cancer
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Stage I or Stage II Non-Small Cell Lung Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0618; CDR0000571744
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT (Experimental): Stereotactic body radiation therapy (SBRT)
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT delivered in 3 fractions of 20 Gy/fraction over 1.5 to 2 weeks for a total of 60 Gy
  Other Names: Stereotactic body radiation therapy; Stereotactic ablative radiotherapy; SABR

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue near the tumor.

PURPOSE: This phase II trial is studying how well stereotactic body radiation therapy works in treating patients with stage I or stage II non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether treatment with radiotherapy involving a high biological dose with limited treatment volume (using stereotactic body radiotherapy [SBRT] techniques) achieves acceptable primary tumor control (i.e., ≥ 90% at 2 years) in patients with resectable early-stage non-small cell lung cancer.

Secondary

* Determine whether treatment with radiotherapy involving a high biological dose with limited treatment volume (using SBRT techniques) achieves acceptable treatment-related toxicity.
* Estimate the disease-free survival and the overall survival rate at 2 years.
* Observe patterns of failure in the first 2 years.
* Assess the level of comorbidity burden on morbidity and efficacy.
* Determine if blood markers prior to, during the course of treatment (between the second and the last dose of SBRT), and at the first follow-up after SBRT predict 2-year primary tumor control and predict for grade ≥ 2 treatment-related toxicities

OUTLINE: This is a multicenter study.

Patients receive 3 fractions of stereotactic body radiotherapy over 14 days. Patients with disease progression undergo surgical resection as salvage local therapy.

After completion of study therapy, patients are followed every 3 months for 2 years, every 6 months for 3 years and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer, including any of the following primary tumor types:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Large cell carcinoma
  * Large cell neuroendocrine tumor
  * Non-small cell carcinoma not otherwise specified
* No pure type bronchoalveolar cell carcinoma
* Stage I or II disease based on 1 of the following combinations of primary tumor, regional nodes, metastasis (TNM) staging:

  * T1, N0, M0
  * T2 (≤ 5 cm), N0, M0
  * T3 (≤ 5 cm), N0, M0 (chest wall primary tumors only)
* No T2 or T3 primary tumors > 5 cm or T3 primary tumors involving the central chest and structures of the mediastinum
* No primary tumor of any T-stage within or touching the zone of the proximal bronchial tree, defined as a volume of 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, or right and left lower lobe bronchi)
* Patients with hilar or mediastinal lymph nodes ≤ 1 cm AND no abnormal hilar or mediastinal uptake on positron emission tomography (PET) scan will be considered N0

  * Patients with > 1 cm hilar or mediastinal lymph nodes on CT scan OR abnormal PET scan (including suspicious but nondiagnostic uptake) will still be eligible if directed tissue biopsies of all abnormally identified areas are negative for cancer
* No direct evidence of regional or distant metastases after appropriate staging studies
* Considered a reasonable candidate for surgical resection of the primary tumor, according to the following criteria:

  * Primary tumor predicted to be technically resectable with a high likelihood of negative surgical margins (as determined by a qualified thoracic surgeon)
  * Baseline forced expiratory volume (FEV)_1 > 35% predicted
  * Postoperative predicted FEV_1 > 30% predicted
  * Diffusion capacity > 35% predicted
  * No hypoxemia (e.g., partial pressure of arterial oxygen (PaO2) of ≤ 60 mm Hg) and/or hypercapnia (e.g., partial pressure of arterial carbon dioxide (PaCO2) > 50 mm Hg) at baseline
  * No severe pulmonary hypertension
  * No severe cerebral, cardiac, or peripheral vascular disease
  * No severe chronic heart disease
* Pleural effusion, if present, must be deemed too small to tap under CT scan guidance and must not be evident on chest x-ray

  * Pleural effusion that appears on chest x-ray will be allowed only after thoracotomy or other invasive procedure

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count ≥ 1,800/mm³
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No synchronous primary or other invasive malignancy within the past 3 years other than nonmelanoma skin cancer or in situ cancer
* No active systemic, pulmonary, or pericardial infection
* No weight loss > 5% for any reason within the past 3 months

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy for lung cancer

  * Prior radiotherapy as part of treatment for head and neck cancer, breast cancer, or other non-lung cancer is allowed provided there will not be significant overlap with the stereotactic body radiotherapy fields
* No prior chemotherapy or surgical resection for this lung cancer
* No other concurrent local or regional antineoplastic therapy (including standard fractionated radiotherapy, non-approved systemic therapy, and surgery), except at disease progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Principal Investigator — Simmons Cancer Center; Elizabeth M. Gore, MD, Study Chair — Medical College of Wisconsin; Harvey I. Pass, MD, Study Chair — NYU Langone Health; Martin J. Edelman, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (19):
- United States (19):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - University of California Davis Cancer Center, Sacramento, California
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - INOVA Alexandria Hospital, Alexandria, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Timmerman RD, Paulus R, Pass HI, Gore EM, Edelman MJ, Galvin J, Straube WL, Nedzi LA, McGarry RC, Robinson CG, Schiff PB, Chang G, Loo BW Jr, Bradley JD, Choy H. Stereotactic Body Radiation Therapy for Operable Early-Stage Lung Cancer: Findings From the NRG Oncology RTOG 0618 Trial. JAMA Oncol. 2018 Sep 1;4(9):1263-1266. doi: 10.1001/jamaoncol.2018.1251. PMID 29852037

RESULTS

PARTICIPANT FLOW:
Groups:
- SBRT: Stereotactic body radiation therapy (SBRT) delivered in 3 fractions of 20 Gy/fraction over 1.5 to 2 weeks for a total of 60 Gy
Period: Overall Study
Arm/Group | SBRT
Started | 33
Completed | 26 (Subjects contributing data to the primary analysis are considered to have completed the study)
Not Completed | 7
Not completed — Protocol Violation | 5
Not completed — Withdrawal by Subject | 1
Not completed — Not treated per protocol and re | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients who started study treatment
Arm/Group | SBRT
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 73 [54 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Primary Tumor Control at 2 Years
Description: Primary tumor control is defined as the absence of primary tumor failure by 2 years after the start of SBRT. Primary tumor failure was considered as the development of either failure within the SBRT treatment fields (in-field failure) or failure within 1.0 cm of the treatment field (marginal failure). An acceptable tumor control rate at 2 years was considered to be 90% (monthly hazard of 0.00439), and an unacceptable rate was 70% (monthly hazard of 0.01486). A one-sided type 1 error of 0.05 and statistical power of 90% was used. A one-sided Z-test was used to determine if the difference between the logarithm of the observed hazard rate and the logarithm of the hypothesized hazard rate of 0.01486 was statistically significant.
Time Frame: From start of treatment to 2 years.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | SBRT
Number analyzed (Participants) | 26
percentage of patients | 96.2 [83.2 to 99.7]

2. Secondary Outcome: Rate of Treatment-related Grade 3 or 4 Toxicity
Description: The development of any treatment-related toxicity from among the following: Gastrointestinal: dysphagia, esophagitis, esophageal stricture/stenosis, esophageal ulceration; Cardiac: pericarditis, pericardial effusion, restrictive cardiomyopathy, ventricular dysfunction (left ventricular diastolic dysfunction, left ventricular systolic dysfunction, right ventricular dysfunction); Neurologic: myelitis, neuropathy (cranial and motor); Hemorrhage: pulmonary or upper respiratory; Pulmonary: decline in pulmonary function as measured by pulmonary function tests (DLCO, FEV1,FVC), pneumonitis, pulmonary fibrosis, hypoxia, pleural effusion, cough, and dyspnea; Any grade 4 or 5 adverse event attributed to the therapy
Time Frame: From start of treatment to end of follow-up. Analysis can occur at or after time of primary outcome measure analysis.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SBRT
Number analyzed (Participants) | 26
percentage of participants | 7.7 [0 to 17.9]

3. Secondary Outcome: Other Grade 3-5 Adverse Events
Description: The development of any treatment-related toxicity not from among the following: Gastrointestinal: dysphagia, esophagitis, esophageal stricture/stenosis, esophageal ulceration; Cardiac: pericarditis, pericardial effusion, restrictive cardiomyopathy, ventricular dysfunction (left ventricular diastolic dysfunction, left ventricular systolic dysfunction, right ventricular dysfunction); Neurologic: myelitis, neuropathy (cranial and motor); Hemorrhage: pulmonary or upper respiratory; Pulmonary: decline in pulmonary function as measured by pulmonary function tests (DLCO, FEV1,FVC), pneumonitis, pulmonary fibrosis, hypoxia, pleural effusion, cough, and dyspnea; Any grade 4 or 5 adverse event attributed to the therapy
Time Frame: From start of treatment to end of follow-up. Analysis can occur at or after time of primary outcome measure analysis.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SBRT
Number analyzed (Participants) | 26
percentage of participants | 3.9 [0 to 19.6]

4. Secondary Outcome: Primary Tumor Failure (PTF), Marginal Failure (MF), Regional Failure (RF), Metastatic Dissemination (MD), Disease-free Survival (DFS), and Overall Survival (OS) at 2 Years
Description: PTF: the development of either failure within the SBRT treatment fields (in-field failure) or failure within 1.0 cm of the treatment field (marginal failure) within the first two years after start of SBRT. RF: the development of measurable tumor within lymph nodes along the natural lymphatic drainage typical for the location of the treated primary disease only with dimension of at least 1.0 cm on imaging studies (preferably CT scans) within the lung, bronchial hilum, or the mediastinum within the first two years after start of SBRT. MD: the appearance after protocol therapy of cancer deposits characteristic of metastatic dissemination from non-small cell lung cancer within the first two years after start of SBRT. DFS: the state of being alive without development of progressive disease, with failure considered the earliest development of either progression or death. OS: the state of being alive, with failure is considered death due to any cause.
Time Frame: From start of treatment to 2 years.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SBRT
Number analyzed (Participants) | 26
percentage of participants
  Primary Tumor Failure at 2 Years | 3.8 [0.3 to 16.8]
  Regional Failure at 2 Years | 7.7 [1.3 to 22.1]
  Metastatic Dissemination at 2 Years | 11.5 [2.8 to 27.1]
  Disease-Free Survival at 2 Years | 73.1 [51.7 to 86.2]
  Overall Survival at 2 Years | 84.6 [64.0 to 93.9]

5. Secondary Outcome: Level of Comorbidity Burden on Morbidity and Efficacy
Time Frame: From start of treatment to end of follow-up.
Population: The data required for this analysis was not obtained and will not be obtained.
Arm/Group | SBRT
Number analyzed (Participants) | 0

6. Secondary Outcome: Assessment of Predictive Value of Blood Markers for Primary Tumor Control at 2 Years and Treatment-related Adverse Events ≥ Grade 2
Description: Assess if blood markers prior to, during the course of treatment (between the second and the last dose of SBRT), and at the first follow-up after SBRT predict 2 year primary tumor control and predict for grade ≥ 2 treatment-related adverse events. Unfortunately, there were not enough specimens submitted to perform this analysis. The specimens that were collected remain in the NRG Oncology Biobank and are available to be combined with other specimens from other studies for an appropriately powered project.
Time Frame: From start of treatment to 2 years.
Population: The data required for this analysis was not obtained and will not be obtained.
Arm/Group | SBRT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | SBRT
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 19/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT (N=26)
Peripheral sensory neuropathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT (N=26)
Chest pain (General disorders) | 2
Fatigue (General disorders) | 2
Pain [other] (General disorders) | 2
Sinusitis [with unknown ANC] (Infections and infestations) | 2
Fracture (Injury, poisoning and procedural complications) | 2
Carbon monoxide diffusing capacity decreased (Investigations) | 13
Forced expiratory volume decreased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3
Joint pain (Musculoskeletal and connective tissue disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 8
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.